CLINICAL TRIAL: NCT01178593
Title: GUT-FOCUSED GROUP HYPNOSIS FOR TREATMENT OF IRRITABLE BOWEL SYNDROME - A RANDOMISED CONTROLLED TRIAL
Brief Title: Group Hypnosis for Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gabriele Moser, ao.Univ.Prof.Dr.med., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FA716E0126
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; RCT; psychology; hypnosis; psychotherapy; group therapy
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Medical Therapy (SMT) (No Intervention): standard medical treatment (care as usual) with supportive talks
- Gut focused hypnotherapy (Active Comparator): weekly sessions of gut focused hypnotherapy in groups (10 sessions within 12 weeks)
  Interventions: Other: Gut-focused hypnotherapy in group sessions

INTERVENTIONS:
Other: Gut-focused hypnotherapy in group sessions — weekly session (45 min) of gut focused hypnotherapy (10 sessions within 12 weeks)
  Other Names: hypnosis; gut directed hypnosis; gut directed hypnotherapy; gut focused hypnosis
  Arms: Gut focused hypnotherapy

SUMMARY:
This randomised controlled trial (RCT) aimed at assessing the efficacy of hypnotherapy in group sessions (GHT) with a 12-months follow-up.

DETAILED DESCRIPTION:
Method:Patients with IBS, fulfilling Rome III criteria, and aged between 18 and 70, were recruited from the University Hospital of Vienna, from primary care physicians and the Austrian IBS patients' organisation by an information letter with an invitation to participate in this RCT. Patients were invited for an interview at the University hospital to confirm the IBS diagnosis according to the guidelines. Exclusion criteria were: pregnancy, bowel surgery, mental retardation, insufficient knowledge of German, a concomitant severe organic and/or psychiatric disease, and recently indicated treatment with anti-depressants. Anti-depressants at a stable dose for longer than three months were allowed for admission to the study. The time for patients to reach the hospital was not to be longer than one hour. Patients with lactose and fructose intolerance as diagnosed by breath tests were not excluded if they had had an adequate diet over a period of more than three weeks without any change of their IBS symptoms.

Randomisation and therapy If 12 patients fulfilled all inclusion criteria they were randomly assigned to one of the two study arms at a 1:1 ratio. Randomisation was done by using permutated blocks of four in order to provide a balanced allocation. The investigator who generated the randomisation schedule was independent of the rest of the trial (blinded). Randomisation was either to supportive talks and symptomatic (standard) medical treatment (SMT, IBS-symptom-related) according to the guidelines (15-17) or to GHT with SMT. The GHT protocol used was the Manchester protocol of gut-directed hypnotherapy ( ) and consisted of 10 weekly sessions (45 minutes) with six patients per group over a treatment period of 12 weeks. GHT was performed at the University Hospital by two experienced physicians, trained in Manchester (UK). At the first session patients were informed about effects of hypnosis and at the third session subjects were given a compact disc (created by hypnotherapists) for practicing at home on a daily basis (practicing was documented). After an induction of hypnosis by closing the eyes a combination of standard deepening procedures followed. Then suggestions for ego-strengthening, power of self-control and gut-specific relaxation were made with hands on abdomen and visualization of slow, rhythmic waves (water, sea, or river) in pleasant, relaxing situations. The final phase involved imagery to increase one's sense of control and self-efficacy over IBS symptoms. GHT patients received also SMT. For control patients the same frequency and duration (45 minutes, SMT) of doctor's visits were offered at the University Hospital provided by a physician with additional qualification in psychosomatic medicine. No kind of relaxation techniques was allowed for control patients during the study. Psychotherapies and (changes of) symptomatic medication were allowed for all patients if indicated. If anti-depressants were taken at a stable dose at baseline, no dose reduction or increase was allowed until the six-month follow-up.

All data were collected by study coordinators not involved in the treatment. Data were entered into SPSS 17.0 and analysed by an independent person with no information about patients' randomisation (blinded).

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS, fulfilling Rome III criteria, and aged between 18 and 70, The time for patients to reach the hospital should not to be longer than one hour

Exclusion Criteria:

pregnancy, bowel surgery, mental retardation, insufficient knowledge of German, a concomitant severe organic and/or psychiatric disease, recently indicated treatment with anti-depressants.-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome - Impact Scale, IBS-IS | May 2008-September 2010
  the IBS-Impact-Scale (IBS-IS). The IBS-IS is a disease-specific documentation of the impact of IBS on patients' lives and was developed and validated for use in clinical trials

SECONDARY OUTCOMES:
Short-Form 36 (SF-36) | May 2008-September 2010
  conveys eight dimensions of Quality of life (QOL): limitations in physical functioning, role limitation due to physical health problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional limitations and mental health (higher scores indicating higher QOL). Validity and reliability have been proven extensively for diverse patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Moser, ao. Prof., Principal Investigator — Medical University of Vienna